CLINICAL TRIAL: NCT04378816
Title: A Patient-centered Continuous and Interdisciplinary Shared Decision Making Approach for Breast Cancer Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: N201912134
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-05

CONDITIONS: Shared Decision Making; Self-Efficacy for Decision Making
Keywords: breast cancer; shared decision making; patient decision aid; question prompt list
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QPL intervention group (Experimental): Using shared decision making support tool(Question Prompt List) for intervention
  Interventions: Other: Shared decision making support tool
- Usual care group (No Intervention): No intervention, just continue using usual care

INTERVENTIONS:
Other: Shared decision making support tool — Health education materials containing treatments and questions about patient values to help patients make the most appropriate decisions.A question prompt list (QPL) is a structured list of questions that serves as a prompt for patients to consider questions to ask their physician.
  Arms: QPL intervention group

SUMMARY:
Background: Breast cancer rehabilitation has gradually expanded from post-surgery rehabilitation to continuous rehabilitation including prehabilitation between cancer diagnosis and surgical treatment, post-surgery rehabilitation, and return-to-work/return-home interventions. Continuous rehabilitation provides patients with tailored training at each treatment period, in order to maintain patients' functions or accelerate the recovery of functions, reduce the burden of symptoms, and improve patients' independence and quality of life. As the functional rehabilitation needs and lifestyle adjustment needs of each patient's life role are different, only with an interprofessional rehabilitation team, patients can obtain patient-centered and comprehensive rehabilitation interventions. Interprofessional shared decision making (IP-SDM) is an decision-making process that interprofessional team and patients discussion the treatment options, based on the best evidence and patient values and preferences, to make a patient-centered treatment decision. However, the major barriers of the implementation of IP-SDM are the lack of IP-SDM skills of clinicians and the lack of medical knowledge of patients.

Purposes: The project aims (1) to develop a patient-centered continuous and interdisciplinary shared decision making approach for breast cancer rehabilitation, including IP-SDM training for interprofessional rehabilitation team, as well as decision coaching, patient decision aid and question prompt list for patients; and (2) to examine the effects of IP-SDM approach on the IP-SDM self-efficacy of interprofessional rehabilitation team and patients, quality of IP-SDM process, patients' satisfaction with decision, concordance between preferences and the chosen options, patients' upper limb function and health-related quality of life.

DETAILED DESCRIPTION:
Methods: This 3-year prospective project will be divided into four phases: (1) Exploration of the IP-SDM needs of continuous breast cancer rehabilitation: We will interview breast cancer patients and consult breast cancer care professionals with different disciplines to understand the IP-SDM needs of breast cancer rehabilitation in each treatment period. (2) Development of communication and decision aids: An expert panel will develop a mobile application prototype of communication and decision aids. The prototype will be testes for the understandability and applicability by breast cancer patients. (3) Development of decision coaching and IP-SDM training programs: We will consult experts to develop a decision coaching training program for breast cancer patients and an IP-SDM training program for interprofessional rehabilitation team. (4) Evaluation of the effectiveness of the patient-centered continuous and interdisciplinary shared decision making approach for breast cancer rehabilitation: We will conduct a parallel-group, single-blinded randomized controlled trial and recruit 116 breast cancer patients at Taipei Medical University Hospital to evaluate the effectiveness of the IP-SDM approach.

Expected results and impacts: We expect that the patient-centered continuous and interdisciplinary shared decision making approach for breast cancer rehabilitation will effectively improve patients' IP-SDM self-efficacy, quality of IP-SDM process, patients' satisfaction with decision, concordance between preferences and the chosen options, patients' upper limb function and health-related quality of life. In the future, this IP-SDM approach will be promising to be applied to other medical institutions and other cancer populations, so as to enhance patient-centered, interprofessional and continuous practice in cancer care.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Breast cancer ICD-10 codes C50、C79.2、C79.81、D05.00-D05.92、D48.60-D48.62、Z51.0、Z51.11; ICD-9 codes 174.0~174.9、198.2、198.81、233.0、238.3、V58.0、V58.1)
* Age>20 years
* Ability to follow instructions and complete the interviews
* Agree to record the doctor-patient communication process

Exclusion Criteria:

* Diagnoses mental problems
* Patient with Cancer terminal stage and weakness
* Cancer has brain metastases or other major diseases (such as dementia) that may affect cognitive function.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-05-05 (Actual); Primary Completion 2021-05-05 (Estimated); Study Completion 2021-05-05 (Estimated)

PRIMARY OUTCOMES:
Control Preference Scale | After intervention immediately
  Control Preference Scale (CPS) is to measure the patients' preferred role whether change in making decisions with the medical provider before intervention and after intervention. It consists of five cards, each of which presents a different character in medical decision-making in a cartoon pattern, and performs a series of comparisons to rank the preference.
Patient-Physician Interactions Questionnaire | After intervention immediately
  Patient-Physician Interactions Questionnaire (PEPPI) is to measure patients' self-efficacy in obtaining medical information and attention to their medical concerns from physicians. It has 10 items and higher scores means self-efficacy performance.
Decision Self Efficacy Scale | After intervention immediately
  Decision Self Efficacy Scale (DSES) is to measure patients' self-confidence and belief in measuring the ability of patients to participate in decision-making. It has 11 items with 5 level Likert scale. The scale range is 0-100 and higher scores indicate better decision self-efficacy.
Patients' Perceived Involvement in Care Scale | After intervention immediately
  Patients' Perceived Involvement in Care Scale (PICS) is to measure three relatively distinct factors: (1) doctor facilitation of patient involvement, (2) level of information exchange, and (3) patient participation in decision making. It has 13 items.

SECONDARY OUTCOMES:
modified brief version of the Health Care Climate Questionnaire | After intervention immediately
  modified brief version of the Health Care Climate Questionnaire (mHCCQ) is to measure patient perceptions of their clinician's autonomy supportive communication. It has 6 items and higher scores means autonomy support performance.
SURE test | After intervention immediately
  SURE test is to measure: (1) certainty about the decision, (2) knowledge of benefits and risks of each option, (3) personal values for benefits and risks, and (4) support and advice to make a choice.11 . It has 6 items and higher score on the SURE test indicates low decisional conflict
State-Trait Anxiety Inventory | After intervention immediately
  State-Trait Anxiety Inventory (STAI) is to measure the level of trait and state anxiety . It has 20 items.
collaboRATE | After intervention immediately
  collaboRATE is to measure the level of shared decision making in the clinical encounter from the patient's perspective is an important part of assessing health care quality and provider performance.It has 3 items.

CONTACTS AND LOCATIONS:
Overall Officials: WEN-HSUAN HOU, Study Director — Taipei Medical University
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No